CLINICAL TRIAL: NCT02072005
Title: Mobile Application Based Personalized Solutions and Tools for Medication Adherence of Rx Pills
Brief Title: Mobile App Based Personalized Solutions and Tools for Medication Adherence of Rx Pills
Acronym: mSMART
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Intelligent Automation, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00048974; HHSN271201300022C (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2014-02-21; First posted 2014-02-26 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Regular cigarette smokers
  Interventions: Other: mSMART smartphone application

INTERVENTIONS:
Other: mSMART smartphone application — This application is an interface that provides subjects with information and questionnaires related to their medication.

SUMMARY:
The primary aim of this study is to conduct a 9-patient feasibility and acceptability study of mSMART (with future studies focusing on improved medication adherence). The sample will include daily smokers who are already taking a prescribed medication. There will be no change in any medication regimen in this study, and the sample will include smokers either with or without a psychiatric disorder. Subjects will be asked to use a smartphone application, or "app" (i.e. mSMART) that will provide information about their medication and when to take it. Along with smart phone, the participants will be asked to utilize an electronic pillbox (i.e. GlowCap) to further assist with medication compliance.

DETAILED DESCRIPTION:
Subjects will be 9 nicotine dependent male and female smokers who take at least one prescribed medication regularly. This sample will allow for psychiatric comorbidity, though is not required. They will be asked to carry a smartphone for 7 days and use a smartphone application, also called an "app," (i.e. mSMART) that will provide information about their medication and when to take it. Along with smart phone, the participants will be asked to utilize an electronic pillbox (i.e. GlowCap) to further assist with medication compliance. The study consists of a Screening Visit (~4½ hours), Training Visit (~1 hour), and 1 Follow-Up Session (~2 hours). Post the Training visit, subjects will then complete the week observation period. During that time, subjects will complete experimenter-prompted assessments to assess factors that may interfere with medication adherence (e.g., psychiatric symptoms, such as forgetfulness). As part of the 'app', reminders will be sent to subjects to take their medication (e.g., the reminders will be programmed to accommodate multiple times a day dosing within dosage schedule windows). Subjects will also be provided with an electronic pillbox that will dispense the subject's medication over the 7 day observation period. After the 7 day period, subjects will return the smartphone at the follow-up visit. Primary outcome variable measured will be medication adherence as an indicator of feasibility and acceptability of the mSMART app.

This study is an observational study since participants will already be taking a medication prescribed by their own physician. The sample is a non-treatment seeking sample of adult cigarette smokers. Participants will not be asked to modify their smoking behavior or medication use in any way. Participants will receive two devices (i.e., [1] the smartphone with mSMART and [2] GlowCap) over the seven day observation period of smoking behavior and medication adherence. The ultimate goal of mSMART is to assist with medication adherence and is thus an intervention, although the goal of this study is to assess how acceptable and feasible it is in a sample already adherent to their medications. We do not predict any changes in smoking behavior or medication adherence once participants are provided with mSMART or GlowCap. GlowCap is being used to allow the investigators to measure times at which the medications were taken.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Male or female
* Taking a prescribed psychiatric or smoking cessation medication in pill form over the past 30 days
* Self-report smoking at least 5 cigarettes/day
* Provides an afternoon exhaled carbon monoxide reading of at least 5 ppm.
* Cognitive functioning > 80 as assessed by the Kaufmann Brief Intelligence Test, second edition (KBIT-II)

Exclusion Criteria:

* Significant and chronic medical problems
* Estimated IQ < 80 on Kaufmann Brief Intelligence Test, Second Edition
* Meets criteria for any other Axis I Disorder (determined by the Structured Diagnostic Interview for DSM; SCID) that requires intervention and might interfere with study participation
* Current non-nicotine substance abuse or dependence or history within the last 3 months
* Females who are pregnant or attempting to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be 15 adult, nicotine dependent smokers for a target completion sample of 9. Subjects will be allowed to meet criteria for a current comorbid psychiatric disorder (e.g., Attention-Deficit/Hyperactivity Disorder [ADHD], Post-Traumatic Stress Disorder, Major Depressive Disorder), though non-psychiatric smokers will be included as well. Participants will be taking some form of prescribed psychiatric medication or nicotine replacement therapy in pill form.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of alarms emitted by msmart app that subjects respond to. | 7 days
  Measurement of app feasibility.
Likert response score | After 7 day observation period.
  Likert scale responses to a questionnaire completed at follow-up visit. Questionnaire asks for agreement with statements relating to acceptability of the app.
  Scale:
  1. = not at all
  2. = somewhat
  3. = moderately
  4. = extremely (example question: What was your overall satisfaction with mSMART?)

SECONDARY OUTCOMES:
Percentage of study participant attrition. | 7 days
  Used to assess acceptability of mSMART app.

CONTACTS AND LOCATIONS:
Overall Officials: John T Mitchell, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States